CLINICAL TRIAL: NCT01049698
Title: Improving Muscle for Functional Independence Trial
Acronym: I'MFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00009098
Record Dates: First submitted 2010-01-11; First posted 2010-01-14 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Older adults; resistance training; exercise
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Resistance Training; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Resistance Training (Active Comparator): 3 d/wk resistance training
  Interventions: Behavioral: Resistance Training
- 2. Resistance Training + Diet (Experimental): Resistance training plus caloric restriction
  Interventions: Behavioral: Resistance Training + Diet

INTERVENTIONS:
Behavioral: Resistance Training — 3 d/wk resistance training
  Other Names: RT; Nautilus resistance machines
  Arms: 1. Resistance Training
Behavioral: Resistance Training + Diet — 3 d/w resistance training plus 600 kcal/d deficit
  Other Names: RT+CR
  Arms: 2. Resistance Training + Diet

SUMMARY:
Aging is associated with declines in muscle strength, power, and overall functional ability that lead to disability and loss of independence. Furthermore, the existing high prevalence of obesity in the elderly is greatly exacerbating these aging-related declines in function. To date, regular exercise, especially resistance exercise, is the only known treatment to consistently improve muscle function and perhaps delay the onset of disability. However, not all individuals experience the same magnitude of benefit from a given exercise stimulus, and accumulating data show that obesity limits muscle adaptations to chronic exercise.Therefore, the proposed study is designed to determine the effects of caloric restriction on improvements in skeletal muscle function in response to RT.

DETAILED DESCRIPTION:
Design Overview:

This is a 5-month randomized trial in 130 older, overweight or obese, sedentary men and women. Phase 1 involves recruitment and screening followed by baseline research testing (Phase 2). Next, subjects will be randomly assigned to one of two 5-month treatments (Phase 3): RT intervention alone (RT) or to an RT with caloric restriction (RT+CR) intervention. Subjects will return for visits the completion of their 5 month intervention. A subset of participants (n=30) will return for an 18 month follow up.

Interventions:

Resistance training+ Caloric Restriction:Participants assigned to RT+CR group will be instructed to follow a hypocaloric diet (-600 kcal/d) for 20 weeks, as well as the resistance training program noted below.In addition, all participants will be provided with a daily calcium (1200 mg/d) and vitamin D (800 IU/d) supplement.The intervention will incorporate meal replacements, nutrition education, and lifestyle behavior modifications.

Resistance training: The maximal weight that can be lifted with correct form in a single repetition (1RM) will be used to prescribe intensity. Strength testing will be repeated every 4 wks and the training loads adjusted so that they are consistent with the 70% 1RM goal. Participants will exercise 3 d/wk on Nautilus resistance machines, under the supervision of two exercise leaders who are trained in basic life support and in emergency management procedures. All exercise will take place at Wake Forest University's Department of Health and Exercise Science Clinical Research Center (CRC). Participants will exercise in small groups which will allow a rotation/rest between machines and enhance the social environment. Heart rate and blood pressure will be measured before and after each session. Subjects will warm-up by walking or cycling for 5 minutes at a slow pace followed by large muscle flexibility exercises. The interventionists will ensure that participants adjust the equipment appropriate to their body size and complete the exercises with correct form. Training sessions will end with a cool-down by walking or cycling for 5 minutes at a slow pace followed by light stretching.

ELIGIBILITY:
Inclusion Criteria:

* BMI=27-34.9 kg/m2
* No resistance training for past 6 mos
* Normal cognitive function (MMSE >24)
* No contraindications for participation in weight loss or resistance exercise including severe arthritis or musculoskeletal disorders, knee or hip replacement or spinal surgery in past year
* No broken bones in the past 6 months
* Able to provide own transportation to study visits and intervention
* Not involved in any other research study and not undergoing physical therapy
* Not dependent on a cane or walker

Exclusion Criteria:

* Weight loss or gain (±5%) in past 6 months
* Body mass >136 kg (DXA limit)
* Current smoker (No nicotine within past year) or evidence of alcohol or drug abuse
* Insulin dependent or uncontrolled diabetes (FBG >140 mg/dL)
* Uncontrolled hypertension (BP>180/100 mmHg)
* Abnormal kidney function or liver blood tests
* Past or current cardiovascular disease, including uncontrolled angina or dysrhythmia, hypertrophic cardiomyopathy, congestive heart failure, PAD, stroke, history of myocardial infarction, use of defibrillator or major heart surgery, or deep vein thrombosis or pulmonary embolus
* Past or current respiratory disease (requiring steroid treatment or supplemental oxygen)
* Past or current clinical diagnoses of neurological or hematological disease
* Use of any medications that could influence study variables (growth/steroid hormones, prescription anti-inflammatory medications, or beta blockers, Coumadin or any other blood thinner, including Plavix, Ticid, and Aggrenox)
* Cancer requiring treatment in past 2 years, except non-melanoma skin cancers
* Clinically evident edema or anemia

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle function (muscle quality and muscle power) and overall physical function (SPPB score) | 5 month study with baseline and 5 and 18 month follow up assessment visits

SECONDARY OUTCOMES:
single-fiber contractile force and power, intramyocellular lipid (IMCL), muscle gene and protein expression of interleukin-6 (IL-6) and tumor necrosis factor alpha. | baseline and 5 and 18-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Nicklas, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available upon email request to the study PI and upon completion of a data-sharing agreement. This agreement will require that data be used only for research purposes, that no attempts be made to identify individual patients, that the data will be kept secure, that the user will not distribute the data to other researchers, that the user will return the files or destroy them once the project is completed, and that the user will acknowledge the data source. All data files will be de-identified. In addition, variables that could permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects will be removed or recoded. We will create a link on our website that describes our study and the data available for data sharing with descriptions.

REFERENCES:
- [Derived] Bharadwaj MS, Tyrrell DJ, Leng I, Demons JL, Lyles MF, Carr JJ, Nicklas BJ, Molina AJ. Relationships between mitochondrial content and bioenergetics with obesity, body composition and fat distribution in healthy older adults. BMC Obes. 2015 Oct 6;2:40. doi: 10.1186/s40608-015-0070-4. eCollection 2015. PMID 26448868
- [Derived] Jefferson ME, Nicklas BJ, Chmelo EA, Crotts CI, Shaltout HA, Diz DI, Marsh AP, Brinkley TE. Effects of Resistance Training With and Without Caloric Restriction on Arterial Stiffness in Overweight and Obese Older Adults. Am J Hypertens. 2016 Apr;29(4):494-500. doi: 10.1093/ajh/hpv139. Epub 2015 Aug 20. PMID 26297029
- [Derived] Nicklas BJ, Chmelo E, Delbono O, Carr JJ, Lyles MF, Marsh AP. Effects of resistance training with and without caloric restriction on physical function and mobility in overweight and obese older adults: a randomized controlled trial. Am J Clin Nutr. 2015 May;101(5):991-9. doi: 10.3945/ajcn.114.105270. Epub 2015 Mar 11. PMID 25762810